CLINICAL TRIAL: NCT04247009
Title: Postprandial Inflammation in Rheumatoid Arthritis
Acronym: PIRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Sahlgrenska University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PIRA
Record Dates: First submitted 2020-01-21; First posted 2020-01-29 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Arthritis, Rheumatoid; Inflammatory Response; Dietary Exposure; Diet, Healthy
Keywords: postprandial; inflammation; rheumatoid arthritis; RA; diet; PIRA
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation | interventions — Fish Products

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All data will be given a new code Before statistical analysis to mask treatment (study meal or Control) to the outcome assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Meat (Active Comparator): Patients with RA served a meal of meat
  Interventions: Other: Meal based on red meat, fish products or vegan products; Other: Meal based on red meat
- Fish (Active Comparator): Patients with RA served a meal of fish
  Interventions: Other: Meal based on red meat, fish products or vegan products
- Vegan (Active Comparator): Patients with RA served a vegan meal
  Interventions: Other: Meal based on red meat, fish products or vegan products
- Meat controls (Active Comparator): Matched controls served a meal of meat
  Interventions: Other: Meal based on red meat

INTERVENTIONS:
Other: Meal based on red meat, fish products or vegan products — Three meals will be served
  Arms: Fish; Meat; Vegan
Other: Meal based on red meat — Matched Controls will be served only one meal of meat to compare response between (non-RA) matched controls and patients with RA
  Arms: Meat; Meat controls

SUMMARY:
Patients with RA will be studied to see whether meals of different content will affect inflammation and metabolic variables in the postprandial state. Healthy controls will also be invited to examine potentially different responses to patients with RA.

DETAILED DESCRIPTION:
The PIRA study aims to evaluate the metabolic and inflammatory effects after a vegan meal or a meal containing red meat or fish in patients with RA and matched controls. The study have a cross-over design and each participant will have one of three meals every week and then be compared to themselves. In addition healthy individuals will be included for the red meat meal so that the response from this meal could be compared between patients with RA and their matched controls. Blood samples will be collected before the meal (fasting) and every hour until 5h. Primary outcome will be high sensitive IL-6. Secondary outcomes will be additional inflammation markers such as area under curve for hs-CRP and gene expression in PBMC:s regarding genes related to inflammation and, glucose, blood lipids and metabolomics-profile in serum and urine.

ELIGIBILITY:
Inclusion Criteria for patients with RA:

* Diagnosed with rheumatoid arthritis
* BMI 18.5-30.0 kg/m2
* 2 years or more since diagnosis
* No DMARD changes during the last 3 months

Inclusion Criteria for healthy controls:

* Absence of diagnosis of RA
* BMI 18.5-30.0 kg/m2
* Self-assessed as healthy

Exclusion Criteria:

* Diagnosis of cancer, inflammatory bowel disease, celiac disease, diabetes
* Allergy or intolerance to any of the foods in the study
* Pregnancy or breastfeeding
* Use of any blood lipid lowering medication, glucocorticoids or IL-6-inhibitor during the last 4 weeks prior to enrolment
* Smoking
* Hemoglobin < 100 g/L

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Circulating interleukin 6 | From baseline up to 5 hours postprandial
  Changes from fasting to postprandial
Circulating high sensitive C-reactive protein (CRP) | From baseline up to 5 hours postprandial
  Changes from fasting to 5 hours postprandial, area under curve
Circulating triacylglycerides | From baseline up to 5 hours postprandial
  Blood lipid levels, Area Under curve from fasting to 5 hours postprandial
Gene expression analysis | From baseline up to 5 hours postprandial
  Changes in gene expressions related to inflammation and disease activity in peripheral blood mononuclear cells
Serum metabolomics | From baseline up to 5 hours postprandial
  Patterns of nuclear magnetic resonance (NMR) analysis of metabolites, analysis of several timepoints separately
Urine metabolomics | From baseline up to 5 hours postprandial
  Patterns of nuclear magnetic resonance (NMR) analysis of metabolites,analysis of several timepoints separately

SECONDARY OUTCOMES:
Body composition | Measured at inclusion of trial, expected to be complete within 6 months
  Measured by dual energy X-ray technology
Body composition | Measured at inclusion and during trial, expected to be complete within 1 year
  measured by electric impedance analysis
Resting metabolic rate | through study completion, expected within 1 year
  measured by indirect calorimetry
Glucose | From baseline up to 5 hours postprandial
  blood glucose levels measured by NMR-analysis
Insulin | From baseline up to 5 hours postprandial
  blood insulin levels measured by NMR-analysis
Patient-reported quality of life | through study completion, expected to be complete within 1 year
  Measured by EQ5D-5L questionnaire
Patient-reported health | through study completion, expected to be complete within 1 year
  Measured by the Short Form (SF36) questionnaire
Patient-reported dietary intake | Through study completion, expected to be complete within 1 year
  measured by food frequency questionnaire and 4-day food diary
Patient-reported background and dietary habits | During trial, expected to be complete within 1 year
  Measured by questionnaire about socioeconomic status and changes in dietary habits related to perceived health
Patient-reported disability | During trial, expected to be complete within 1 year
  Health Assessment Questionnaire, disability index (HAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Helen HL Lindqvist, PhD, Principal Investigator — Göteborg University
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Not in US/Canada, Sweden

IPD SHARING:
Plan to Share IPD: No
Data cannot be shared publicly because of Swedish law. The datasets analysed could be made available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Lindqvist HM, Hulander E, Barebring L, Gjertsson I, Winkvist A. A randomized controlled cross-over trial of differences in acute effects on serum metabolites from isocaloric meals based on red meat, fatty fish, or soy protein. Eur J Nutr. 2025 May 26;64(5):187. doi: 10.1007/s00394-025-03710-0. PMID 40418340
- [Derived] Sallstrom T, Barebring L, Hulander E, Gjertsson I, Winkvist A, Lindqvist HM. Inflammatory and lipemic response to red meat intake in women with and without Rheumatoid Arthritis: a single meal study within a randomized controlled trial. BMC Nutr. 2025 Apr 11;11(1):74. doi: 10.1186/s40795-025-01055-9. PMID 40217385
- [Derived] Lindqvist HM, Gjertsson I, Hulander E, Barebring L, Winkvist A. Exploring the differences in serum metabolite profiles after intake of red meat in women with rheumatoid arthritis and a matched control group. Eur J Nutr. 2024 Feb;63(1):221-230. doi: 10.1007/s00394-023-03257-y. Epub 2023 Oct 9. PMID 37814020
- [Derived] Lindqvist HM, Wallengren O, Eriksson A, Hulander E, Winkvist A, Barebring L. Validity of bioimpedance for assessment of fat-free mass in women with Rheumatoid Arthritis compared to non-rheumatic controls. Clin Nutr ESPEN. 2022 Feb;47:333-338. doi: 10.1016/j.clnesp.2021.11.016. Epub 2021 Nov 14. PMID 35063223